CLINICAL TRIAL: NCT05671120
Title: Transcutaneous Levator Recession for Non-thyroid Lid Retraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ehab tharwat, Principal investigator, Al-Azhar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: levator recession
Record Dates: First submitted 2023-01-01; First posted 2023-01-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Eye Diseases
MeSH Terms: conditions — Eye Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transcutaneous levator recession (Other)
  Interventions: Procedure: Transcutaneous levator recession

INTERVENTIONS:
Procedure: Transcutaneous levator recession — recession of the upper and lower eyelid retractors can improve the upper eyelid contour if the patient has lateral flare (common in TED). The choice of procedure depends on severity of lid retraction and associated features like proptosis, status of extraocular muscles, and corneal condition

SUMMARY:
This work aims to describe and assess the efficacy of transcutaneous levator palpebrea superioris muscle recession as a surgical procedure for treatment of upper lid retraction of various causes other than thyroid eye disease

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from upper eyelid retraction of various causes other than thyroid eye disease

Exclusion Criteria:

* Patients refused to participate in the study, patients with systemic diseases causing lid retraction (such as Guillain-Barré syndrome), pseudo retractions, contralateral ptosis, local skin condition (as scar adherence), medication (such as sympathomimetic drugs, lithium, and steroid), neurological conditions (such as dorsal midbrain syndrome and hydrocephalus) and thyroid related lid retraction

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-08-02 (Actual)

PRIMARY OUTCOMES:
Margin reflex distance (MRD1) | Baseline
  MRD1 is a commonly used parameter in the assessment of patients with blepharoptosis and is defined as the distance between the upper lid margin and the corneal reflex when the eye is in the primary position
Margin reflex distance (MRD1) | at one month post operative
  MRD1 is a commonly used parameter in the assessment of patients with blepharoptosis and is defined as the distance between the upper lid margin and the corneal reflex when the eye is in the primary position

CONTACTS AND LOCATIONS:
Locations (1):
- Ehab tharwat, Damietta, New Damietta, Egypt

IPD SHARING:
Plan to Share IPD: No